CLINICAL TRIAL: NCT00833768
Title: A Randomised, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Sevelamer Carbonate Tablets Dosed Three Times a Day in Hyperphosphataemic Chronic Kidney Disease (CKD) Patients Not on Dialysis
Brief Title: A Randomised, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Sevelamer Carbonate Tablets Dosed Three Times a Day in Hyperphosphataemic Chronic Kidney Disease Patients Not on Dialysis
Acronym: ASPIRE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: After an extensive review,the ASPIRE in CKD study was terminated because it was not possible to complete the study in an appropriate time frame.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SVCARB00606; Eudra CT: 2007-003885-16 (Registry Identifier: EudraCT)
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Kidney Disease; Hyperphosphatemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — Sevelamer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevelamer carbonate (Active Comparator)
  Interventions: Drug: Sevelamer carbonate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo for sevelamer carbonate

INTERVENTIONS:
Drug: Sevelamer carbonate — 800mg tablets to be taken orally with meals three times per day
  Other Names: Renvela(TM)
  Arms: Sevelamer carbonate
Drug: Placebo for sevelamer carbonate — Placebo tablets to be taken orally with meals three times per day
  Arms: Placebo

SUMMARY:
Approximately 207 hyperphosphatemic CKD patients not on dialysis will be entered into this study at approximately 50 sites within approximately 9 European countries. The purpose of this study is to determine if sevelamer carbonate tablets dosed three times a day (TID) is a safe and effective treatment for the control of serum phosphorous levels in hyperphosphatemic CKD patients not on dialysis. Total length of participation is approximately 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Serum phosphorus measurement ≥4.6 mg/dL (≥1.49 mmol/L) and ≤5.5 mg/dL (≤1.76 mmol/L after discontinuation of current phosphate binder therapy if applicable.

Exclusion Criteria:

* Active dysphagia or swallowing disorder or a predisposition to or current bowel obstruction, ileus, or severe gastrointestinal motility disorders including severe constipation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy and safety of sevelamer carbonate and placebo dosed three times per day (TID) on serum phosphorus levels | 24 weeks

SECONDARY OUTCOMES:
To compare the efficacy and safety of sevelamer carbonate and placebo dosed three times per day (TID) on serum total cholesterol and low density lipoprotein (LDL) cholesterol | 24 weeks
To compare the efficacy and safety of sevelamer carbonate and placebo dosed three times per day (TID) on serum corrected calcium-phosphorus product (CaxP) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (36):
- Austria (4):
  - Universitätsklinik für Innere Medizin, Klinische Abteilung für Nephrologie und Hämodialyse, Graz
  - Uniklinik für Innere Medizin IV, Nephrologie und Hypertensiologie, Zentrum für Innere Medizin, Medizinische Universität Innsbruck, Innsbruck
  - Krankenhaus der Elisabethinen Linz, 3. Abteilung Schwerpunkt Nephrologie, Linz
  - Universitätsklinik für Innere Medizin III, Klinische Abteilung für Nephrologie und Dialyse, Vienna
- France (7):
  - CHU Amiens Sud Service de Néphrologie, Amiens
  - Hôpital Pellegrin Service de Néphrologie, Bordeaux
  - Hôpital Européen G. Pompidou Département de Physiologie - Explorations Fonctionnelles et Radio-Isotopes, Cedex
  - Service de Néphrologie Hémodialyse Clinique de l'Orangerie, Cedex
  - Hôpital La Peyronie Nephrologie, Montpellier
  - Hôpital Tenon Néphrologie Hémodialyse, Paris
  - CHU de Brabois, Service de Néphrologie, Vandœuvre-lès-Nancy
- Germany (3):
  - Klinikum Darmstadt, Darmstadt
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum rechts der Isar der TU München, Nephrologie, München
- Greece (3):
  - Ippokrateio Hospital of Athens, Athens
  - University Hospital of Ioannina, Ioannina
  - General Hospital of Nikaia, Nikaia Peiraias
- Hungary (4):
  - Petz Aladár County Teaching hospital, Department ofimmunonephrology and hypertension, Győr
  - Kaposi Mór County Hospital Department of Nephrology, Kaposvár
  - Szekszárd EuroCare Dialysis Centre Number 7, Szekszárd
  - Kórház u. 1, Veszprém
- Italy (3):
  - Azienda Ospedaliera di Lecco, Lecco
  - Fondazione Salvatore Maugeri, Divisione Nefrologia ed Emodialisi, Pavia
  - Unita' Operativa Complessa Di Nefrologia e Dialisi San Camillo Forlanini, Roma
- Portugal (4):
  - Hospital Santa Cruz, Carnaxide
  - Centro Hospitalar de Coimbra - Serviço de Nefrologia, Coimbra
  - Hospital da Universidade de Coimbra - Serviço de Nefrologia, Av., Coimbra
  - Hospital de São João EPE - Serviço de Nefrologia, Porto
- Spain (5):
  - Servicio de nefrología Fundacion Puigvert, Barcelona
  - Servicio de nefrología H. Arquitecto Marcide, Ferrol
  - Servicio de nefrología Hospital de Galdakao, Galdakao
  - Servicio de nefrología Fundación Hospital Alcorcón, Madrid
  - Servicio de Nefrología, Hospital Universitario Dr Peset,, Valencia
- Sweden (3):
  - Department of Nephrology Sahlgrenska University Hospital, Gothenburg
  - NjurmedicinKliniken Centralsjukhuset, Karlstad
  - Njurmedicinska Kliniken, Karolinska Universitetssjukhuset, Solna, Stockholm